CLINICAL TRIAL: NCT00434369
Title: A Multi-Center, Open-Label, Single-Arm Phase II Trial Assessing the Efficacy and Safety of Weekly Bolus Infusions of 5-Fluorouracil Combined With CoFactor (5-10 Methylenetetrahydrofolate) in Advanced Breast Cancer Patients Who Failed Anthracycline and Taxane Chemotherapy Regimens
Brief Title: 5-Fluorouracil Combined With CoFactor (5-10 Methylenetetrahydrofolate) in Treating Advanced Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mast Therapeutics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 510-08
Record Dates: First submitted 2007-02-07; First posted 2007-02-13 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 5,11-methenyltetrahydrohomofolate

INTERVENTIONS:
Drug: CoFactor (ANX-510)

SUMMARY:
A multi-center, open-label, single-arm Phase II trial assessing the efficacy and safety of weekly bolus infusions of 5-fluorouracil combined with CoFactor (5-10 methylenetetrahydrofolate) in advanced breast cancer patients who failed anthracycline and taxane chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Women with a histologically/cytologically proven diagnosis of advanced adenocarcinoma of the breast.
* Measurable disease. At least one unidimensionally measurable non-bony lesion with a diameter >=10 mm using spiral CT scans (use of spiral CT must be documented in medical records and used consistently throughout the study) or >= 20 mm using conventional CT or MRI scans outside the irradiated area according to RECIST criteria.
* Patients having failed both prior anthracycline and taxane derivative chemotherapy regimens. Anthrocycline and Taxane failure definitions as defined in the protocol.
* No more than two prior chemotherapy regimens for advanced disease.
* Performance status (ECOG) <= 2 or Karnofsky >= 70
* Age >= 18 years.
* Life expectancy >= 12 weeks.
* Adequate organ function as shown by the following:

  1. WBCs >= 3.0 x 109/L, absolute neutrophil count (ANC)>= 1.5 x 109/L, platelets >= 100 x 109/L, hemoglobin >= 9 g/dL
  2. Bilirubin <= 1.25 x the upper limit of normal (ULN),aspartate aminotransferase(AST or alanine aminotransferase(ALT),= 3 x ULN (or <= 5 x ULN in case of liver metastases)
  3. Serum calcium within normal limits
  4. Serum albumin within the normal range for the study site
  5. Creatinine clearance >= 60 mL/min (Cockroft and Gault)
  6. Left ventricular ejection fraction (LVEF) within normal limits as shown by echocardiography or scintigraphy (multiple-gated acquisition scan).
* Patients of childbearing potential must be using medically acceptable contraception for 4 weeks before start of study treatment and 4 months after study treatment completion. Patients of childbearing potential must have a negative pregnancy test result within 7 days prior to study treatment initiation.
* Patients with parenchymal brain metastases must be either adequately controlled following resection or completed appropriate radiation therapy and be receiving a stable corticosteroid dose prior to study entry. Patients with leptomeningeal involvement should not be included in the study.

Exclusion Criteria:

* Her2/neu positive tumor (2+ or 3+).
* Pregnancy or lactation
* Systemic cytotoxic anti-cancer therapy within <=4 weeks of study entry, or 6 weeks if the systemic therapy contains a nitrosourea or mitomycin C. Hormonal anti-cancer treatment must be ongoing, or must have been discontinued >3 months before study entry.
* Prior 5-FU- and/or capecitabine-based palliative chemotherapy.
* Extensive prior radiotherapy affecting more than 30% of bone marrow reserves, or bone marrow / stem cell transplantation.
* Participation in clinical studies of non-approved experimental agents or procedures within <=4 weeks of study entry.
* History of other malignancy, unless cured and the patient has been disease-free for >=2 years. Patients with a history of cervical carcinoma in situ or cured stage I cervical cancer, or of epidermal or basal cell skin cancer, may be eligible for enrollment after discussion with the sponsor.
* Previous unexpected reaction to fluoropyrimidines, with or without documented deficiency of dihydropyrimidine dehydrogenase, or known hypersensitivity to 5-FU.
* Psychologic, familial, sociologic or geographic conditions which do not permit compliance with the study protocol and/or study.
* Significant cardiac disease, including symptomatic ventricular arrhythmia, congestive heart failure, myocardial infarction within 12 months before study entry.
* Concomitant treatment with any experimental drug or anti-cancer drug, except hormone therapy or bisphosphonates.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2006-02

PRIMARY OUTCOMES:
Overall Response Rate

SECONDARY OUTCOMES:
Progression Free Survival
Overall Survival
Duration of Response

CONTACTS AND LOCATIONS:
Locations (6):
- Clinical Research Site in, Buenos Aires, Argentina
- Clinical Investigative Site, Acapulco, Mexico
- Clinical Investigative Site, Lima, Peru
- Russia (2):
  - Clinical Research Site in, Kazan'
  - Clinical Investigative Site, Saint Petersburg
- Clinical Investigative Site, Valencia, Spain